CLINICAL TRIAL: NCT06574438
Title: The Effectiveness of Artificial Intelligence Family Involvement Generative Agent (AIFIGA) Program on Nursing Home Nursing Staff and Family and Residents'Health
Brief Title: The Effectiveness of AIFIGA Program on Nursing Home Nursing Staff and Family and Residents'Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202400678B0
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-06

CONDITIONS: Family; Nursing Home; Digital Health

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIFIGA group (Experimental): receives the AIFIGA program and uses it for 3 months
  Interventions: Behavioral: AIFIGA program
- control group (No Intervention): receives only routine care

INTERVENTIONS:
Behavioral: AIFIGA program — receives the Artificial Intelligence Family Involvement Generative Agent (AIFIGA) program and uses it for 3 months
  Arms: AIFIGA group

SUMMARY:
This study aims to develop and evaluate the longitudinal effectiveness of the Artificial Intelligence Family Involvement Generative Agent (AIFIGA) program in enhancing the health of nursing staff, family, and residents' health through the use of a sequential, mixed methods research design. The development of a real-time, interactive, and informative AIFIGA program that sparks innovation is necessary to achieve effective communication between families and nursing staff.

In Phase I, lasting 18 months, we will develop the AIFIGA program based on triangulate research design, observation and in-depth interview understanding the daily communication experiences and expectations from both families and nursing staff perception in Nursing Homes(NHs) after COVID-19, as well as our previous years' research results. The training data for AIFIGA will be derived from the collection of communication dialogues in these qualitative data. Furthermore, the intelligence of AIFIGA will be developed using publicly available large language models (LLMs).

In Phase II, spanning the next 18 months, we will evaluate the longitudinal effects of the AIFIGA program on the health of residents, families, and nursing staff, tracking changes over time (baseline, 1 month, 3 months, and 6 months). There will be two groups of participants: (a) an AIFIGA group that receives the AIFIGA program and uses it for 3 months, and (b) a control group that receives only routine care.

ELIGIBILITY:
Inclusion Criteria:

All resident-caregiver pairs meeting the inclusion criteria will be invited to join the study.

1. residents aged ≥ 60 years, resident's family were aged equal or higher than 20 years.
2. both residents and family can communicate in Mandarin or Taiwanese
3. residents have a Mini-Mental State Examination (MMSE) score equal to or higher than 16 for residents with no formal education or higher than 24 for residents with at least a primary school education
4. both residents and family agree to participate
5. the family is a significant member of the resident, such as a caregiver.

For nurses and nursing aides:

1. working in the selected nursing home who agree to participate in our program.
2. aged equal or higher than 20 years.

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
resident health-Geriatric Depression Scale (GDS) | baseline, 1 month, 3 months and 6 months
  scale for depression( scored from 0 through to 15.Scores of 0-4 are considered normal; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.)
resident health-Activity of daily living (ADL) | baseline, 1 month, 3 months and 6 months
  assess individual's ability to perform basic self-care tasks (scored from 0 through to 100. higher scores mean more independence)
social support scale | baseline
  Evaluated quantities of social support (four-point Likert scale, where higher scores indicate a greater amount of each type of social resource) & satisfaction with social support (five-point Likert scale, where higher scores indicate greater satisfaction with social support)
brief Center for Epidemiological Studies Depression Scale(CESD-10) | baseline, 1 month, 3 months and 6 months
  assessment for family' depressive status.(scored from 0 through to 30. Any score equal to or above 10 is considered depressed)
The General Health Questionnaire-12(GHQ-12) | baseline, 1 month, 3 months and 6 months
  assessing the mental health status of respondents. ( total score ranges from 0 to 36, Higher scores mean better mental health status outcome)
Family Meaning of Nursing-Home Visits scale | baseline, 1 month, 3 months and 6 months
  measurement of family visiting involvement meaning

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu Hsin Tsai, PhD, Study Chair — Chang Gung University
Locations (1):
- Catholic Mercy Hospital Attached Nursing Home, Hsinchu, Taiwan